CLINICAL TRIAL: NCT00647673
Title: Single-Dose Fasting Bioequivalence Study of Verapamil HCl Extended-Release Capsules (300 mg; Mylan) to Verelan® PM Extended-Release Capsules (300 mg; Schwarz) in Healthy Volunteers Dosed in the Evening
Brief Title: Fasting Study of Verapamil HCl Extended-Release Capsules 300 mg and Verelan® PM Extended-Release Capsules 300 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullivan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: VERA-05134
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy

ARMS (2):
- 1 (Experimental): Verapamil HCL Extended-Release Capsules 300 mg
  Interventions: Drug: Verapamil HCL Extended-Release Capsules 300 mg
- 2 (Active Comparator): Verelan® PM Extended-release Capsules 300 mg
  Interventions: Drug: Verelan® PM Extended-Release Capsules 300 mg

INTERVENTIONS:
Drug: Verapamil HCL Extended-Release Capsules 300 mg — 300mg, single dose fasting
  Arms: 1
Drug: Verelan® PM Extended-Release Capsules 300 mg — 300mg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's verapamil HCl extended-release 300 mg capsules to Schwarz's Verelan® PM extended-release 300 mg capsules following evening administration of a single, oral 300 mg (1 x 300 mg) dose under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Male and/or non-pregnant, non-lactating female.

   1. Women of childbearing potential must have a negative serum (β HCG) pregnancy test performed within 21 days prior to the start of the study and on the evening prior to each dose administration. If dosing is scheduled on Sunday or Monday, serum for β HCG testing may be collected within 48 hours prior to dosing for each study period. An additional serum (β HCG) pregnancy test will be performed upon completion of the study.
   2. Women of childbearing potential must practice abstinence or use an acceptable form of contraception throughout the duration of the study. No hormonal contraceptives or hormonal replacement therapies are permitted in this study. Acceptable forms of contraception include the following:

      1. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
      2. barrier methods containing or used in conjunction with a spermicidal agent, or
      3. surgical sterilization
   3. Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

      1. postmenopausal with an absence of menses for at least one (1) year, or
      2. bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
      3. total hysterectomy
   4. During the course of the study, from study screen until study exit - including the washout period, all men and women of childbearing potential must use a spermicide containing barrier method of contraception in addition to their current contraceptive method. This advice should be documented in the informed consent form.
3. Weight: At least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women and all subjects having a Body Mass Index (BMI) greater than or equal to 19 but less than or equal to 30 (see Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, hepatitis B and hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 21 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within 14 days prior to the initial dose of study medication.
   2. Use of any hormonal contraceptives and hormone replacement therapy within 3 months prior to study medication dosing.
   3. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic disease.
   2. History of any significant cardiovascular disease, including a history of a known accessory bypass tract (Wolff-Parkinson-White or Lown-Ganong-Levine), paroxysmal supraventricular tachycardia, atrial flutter, and hypotension.
   3. Acute illness at the time of either the pre-study medical evaluation or dosing.
   4. A positive HIV, hepatitis B, or hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to verapamil hydrochloride or any other related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Bradycardia less than 50 beats/minute in the supine position, as measured by ECG, at the screening visit or prior to Period I Day 1 dosing.
11. Sitting pulse rate of less than 60 beats per minute and a sitting systolic blood pressure less than 90 or greater than 140 or a sitting diastolic blood pressure less than 60 or greater than 90 after a five-minute resting period at the Screening Visit or prior to Period I Day 1 dosing.
12. Subjects whose diurnal sleep pattern may be altered (i.e., shift workers).
13. Consumption of grapefruit or any grapefruit containing products within 7 days of drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html